CLINICAL TRIAL: NCT03895983
Title: SsST Segment Resolution After Primary Percutaneous Coronary Intervention. A Comparison Between Primary Percutaneous Coronary Intervention With and Without Thrombus Aspiration
Brief Title: ST Segment Resolution After Primary Percutaneous Coronary Intervention.
Acronym: STresolution
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Ragab Abdel mageed, Principal investigator, Assiut University
Other Study IDs: AssiutU37
Record Dates: First submitted 2019-03-24; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombus aspiration group: Will include 135 patients who will have PPCI with thrombus aspiration
  Interventions: Procedure: Percutaneous primary coronary intervention
- Standard PPCI group: Will include 135 patients who will have PPCI without thrombus aspiration
  Interventions: Procedure: Percutaneous primary coronary intervention

INTERVENTIONS:
Procedure: Percutaneous primary coronary intervention — Percutaneous primary coronary intervention

SUMMARY:
To compare the ST segment resolution after primary percutaneous coronary intervention (PPCI) with and without thrombus aspiration in patients with ST segment elevation myocardial infarction as ST segment resolution is the best indicator for the prediction of the outcome and MACE

DETAILED DESCRIPTION:
The idea of an occluding thrombus and its dissolution had been stated since the 1950s.1 Thrombus is present in the infarct-related artery in 88% of patients undergoing coronary artery angiography within the first 4 h of acute myocardial infarction (AMI).

The finding of ST segment elevation in a patient presenting with chest pain allows rapid identification of those who benefit from emergency reperfusion.

Primary percutaneous coronary intervention (PPCI) is now the preferred strategy for emergency reperfusion in patients presenting with ST elevation myocardial infarction (STEMI).

Thrombus aspiration (TA) might be an effective procedure for reducing distal embolization and improving microvascular perfusion in ST-segment elevation myocardial infarction (STEMI), especially in patients with high thrombus burden.

Despite the class III recommendation for routine Thrombus Aspiration use before balloon angioplasty or stenting. manual Thrombus Aspiration might still remain a useful strategy for the interventional cardiologist when treating selected patients with significant thrombus burden during PPCI.

Thrombus grading is classified as:

Grade 0: No angiographic characteristics of thrombus are present. Grade 1: Possible thrombus is present with a such characteristics as: Reduced contrast density, haziness, irregular lesion contour Or smooth convex meniscus at the site of total occlusion Suggestive but not diagnostic of the thrombus.

Grade 2: There is a definite thrombus with greatest dimension <1/2 the vessel diameter.

Grade 3: There is a definite thrombus but with greatest linear dimension>1/2 but <2 vessel dimension.

Grade 4: There is a definite thrombus but with greatest linear dimension >2 vessel dimension.

Grade 5: There is a total occlusion (unable to assess thrombus burden due to total vessel occlusion.

The analysis of ST-segment resolution on the electrocardiogram (ECG) consists of a simple tool, of easy use and low cost, able to document success of the epicardial reperfusion and tissue reperfusion after primary PCI.

The persistence of ST-segment elevation on the ECG, despite the restoration of a normal epicardial flow, signifies a poor prognosis; such persistence is known to be associated with larger infarct size and higher combined rate of severe cardiovascular adverse events.

ELIGIBILITY:
Inclusion Criteria:

. patients with STEMI within 24 hours of chest pain.patients killip class 1 is included in this study

xclusion Criteria:

* killip II-IV
* Previous myocardial infarction
* Patients with left bundle branch block
* Patients with advanced cancer disease
* Patients qith contraindications to anti-coagulation
* Patients with sensitivity to clopidogrel

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 270 patients
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
ST segment resolution | Within 90 minutes after the procedure
  ST segment resolution in relation to the procedure used in primary percutaneous coronary intervention

SECONDARY OUTCOMES:
MACE | one week
  the major adverse coronary events in correlation to ST segment resolution after primary percutaneous coronary intervention (recurrent angina, reinfarction, heart failure, major bleeding, disabling stroke or death) during the period of hospitalization.

IPD SHARING:
Plan to Share IPD: Undecided